CLINICAL TRIAL: NCT00944476
Title: Application of Magnetic Resonance Fat-Free Imaging
Status: Terminated | Type: Observational
Why Stopped: Software issues not resolved.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-078
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Sarcoma
Keywords: Sarcoma; soft tissue; MRI; Questionnaire; 09-078
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pts/volunteers getting regular MRI exam: Fat-free MRI images utilizing standard magnetization transfer imaging will be acquired on 10 patients known or suspected sarcoma of the of the extremity or trunk, in addition to their traditional clinical MRI. In addition, we will perform the same scans on 4 volunteers who have no history of sarcoma.
  Interventions: Procedure: Fat-free MRI images utilizing standard magnetization, Questionnaire before the MRI exam

INTERVENTIONS:
Procedure: Fat-free MRI images utilizing standard magnetization, Questionnaire before the MRI exam — In addition to the traditional MRI exam for clinical use, a fat-free MRI based on standard magnetization transfer magnetic resonance imaging will be acquired. Pts will spend 20 extra minutes and 20 minutes total for volunteers in the MRI scanner. Patients/volunteers will complete the MR Screening Questionnaire before the MRI exam.

SUMMARY:
Magnetic resonance imaging (MRI) is presently the best study for assessing the size and extent of the patient's sarcoma. Many sarcomas contain fat that can interfere with the accuracy of sarcoma detection. The investigators have developed a new MRI method that can suppress all the fat signals in the patient's tumor and this may improve the investigators' ability to see the patient's sarcoma. The purpose of this study is to determine if the investigators' new fat-free imaging methods provides them with images that are better than, equal to, or worse than those images obtained by standard MRI methods. This study may help the investigators develop a more accurate MRI examination.

DETAILED DESCRIPTION:
In addition, we will perform the same scans on 4 volunteers who have no history of sarcoma. Scanning volunteers will allow us to optimize the imaging technique by 1.) Determine the best combination of pulse-sequence and magnetization transfer technique to obtain the greatest contrast and 2.) Determine the parameters of repetition time (TR), echo time (TE) and magnetization transfer time and power in order to reduce overall image acquisition time while optimizing image quality. Honing this technique on volunteers will allow us to decrease scan time and potential discomfort for patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of providing verbal consent.
* 18 years of age or older.
* Participants will belong to one of the following two categories:
* Patient with a known or suspected soft tissue sarcoma of the extremity or trunk who is/will be scheduled for an MRI scan as part of their routine care, -OR--
* Volunteer with no history of sarcoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research participants from those patients who are/will be scheduled for MRI examination as part of their routine clinical care at MSKCC. Dr. Singer will also identify four volunteers with no history of sarcoma to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine if our magnetization transfer fat-free imaging methods produce fat suppression images of sarcoma that are better, equal to or less in quality than fat-suppressed T2-weighted MRI images. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Singer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering CancerCenter, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm